CLINICAL TRIAL: NCT06640543
Title: Effect of Kinesiotape Versus Myofascial Release on Postnatal Low Back Pain: a Randomised Controlled Trial
Brief Title: Effect of Kinesiotape Versus Myofascial Release on Postnatal Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed Mahmoud Ahmed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004348
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Athletic Tape; Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiotape group (Experimental): The participants will be treated with kinesiotape for 4 weeks
  Interventions: Other: Kinesiotape
- myofascial release group (Experimental): The participants will be treated with myofascial release for 4 weeks
  Interventions: Other: Myofascial release

INTERVENTIONS:
Other: Kinesiotape — Postnatal women with low back pain will be treated with kinesiotape, three times per week for 4 weeks
  Arms: kinesiotape group
Other: Myofascial release — Postnatal women with low back pain will be treated with myofascial release for 25 minutes three times per week for 4 weeks
  Arms: myofascial release group

SUMMARY:
This study aims to determine the difference between the effect of kinesiotape and myofascial release in the treatment of postnatal low back pain.

DETAILED DESCRIPTION:
Postpartum back pain may occur in up to 44% of women after childbirth. People who have chronic back pain may have a limited range of motion and/or tenderness upon touch.

Therapeutic KT can benefit a wide variety of musculoskeletal and sports injuries, plus inflammatory conditions. According to the Kinesiotape Method Manual, this traction promotes an elevation of the epidermis and reduces pressure on the mechanoreceptors located below the dermis, thereby reducing nociceptive stimuli and low back pain.

Myofascial release (MFR) is a treatment that uses gentle pressure and stretching to facilitate the release of fascial restrictions caused by accidents, injury, stress, repetitive use, and traumatic or surgical scarring.

Myofascial release is a form of soft tissue therapy used to treat somatic dysfunction and accompanying pain and restriction of motion. This is accomplished by relaxing the contracted muscle, increasing circulation, increasing venous and lymphatic drainage, and stimulating the stretch reflex of muscles and overlying fascia so, reducing low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Their ages will be ranged from 20 to 35 years old.
* Their body mass index (BMI) will not exceed 30 kg/m2.
* Women will be postnatal period by 6-8 weeks.
* All women will be diagnosed by the physician as postnatal low back pain.

Exclusion Criteria:

* Spinal fracture or any other neurological disorders.
* Lumbar disc herniation or degenerative disc disease
* Lumbar spinal stenosis from lumbar disc herniation, degenerative joint disease, or spondylolisthesis
* Women with BMI exceed 30 kg/m2.
* Patients who have polyneuropathy or other neurological disorders.
* Skin disease interferes with kinesiotape or myofascial release application.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity level | 4 weeks
  The intensity of postnatal low back pain will be assessed using a visual analogue scale (VAS) for all participants in both groups before and after treatment, which is a method of representing subjects' pain on a 10 cm linear scale. A score of 0 means " no pain" and 10 means " very high degree of pain

SECONDARY OUTCOMES:
Lumbar flexion range of motion | 4 weeks
  The modified Schober test will be used to measure the lumbar flexion range of motion (ROM) by using the tape measurement. Each participant will be asked to stand erect with her feet about shoulder-width apart to stabilize the pelvis. Then, the posterior superior iliac spines(PSIS) will be determined by the therapist's both thumbs, and then an ink line will be drawn along the midline of the lumbar spines horizontal to the PSIS to mark the midpoint between the two PSIS. Then tape will be used to identify and mark two points: one is 10 cm superior to the midpoint (A), and another is 5 cm inferior to the midpoint (B). The participant will be instructed to bend forward as much as she can while keeping both knees straight, the new distance between superior and inferior skin marking will be measured in centimeters. The increased distance along the tape due to lumbar flexion is normally about 6-7 cm (less than 5 cm should be considered abnormal).
Lumbar extension range of motion | 4 weeks
  The modified Schober test will be used to measure the lumbar extension range of motion (ROM) by using the tape measurement while the patient is in a standing position. The participant will be instructed to put her hands on her buttocks and bend backward into full lumbar extension and the new distance between the superior and inferior skin markings will be measured in centimeters by the tape measurement. The change in the difference between the marks is used to indicate the amount of lumbar extension. The increased distance along the tape due to the extension of the lumbar spine is normally about 2-3 cm (less than 1cm should be considered abnormal).
Lumbar lateral flexion range of motion | 4 weeks
  The participant will be asked to stand erect with her feet about shoulder-width apart. Both right and left lateral flexion will be measured by the tape as the distance from the tip of the index finger to the floor at maximal comfortable lateral flexion. The participant will be instructed to bend her trunk laterally as much as she can. The normal value of lateral spinal flexion is 16.2-28.0 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf M Botla, Professor, Study Director — Cairo University; Mohamed Awad, Professor, Study Chair — Cairo University
Locations (1):
- Mahmoud Ahmed Mahmoud, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol